CLINICAL TRIAL: NCT03520036
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Efficacy, Safety, and Tolerability of MT-7117 in Subjects With Erythropoietic Protoporphyria
Brief Title: Study to Evaluate Efficacy, Safety, and Tolerability of MT-7117 in Subjects With Erythropoietic Protoporphyria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-7117-A01
Record Dates: First submitted 2018-04-23; First posted 2018-05-09 (Actual); Results first posted 2023-01-20 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Erythropoietic Protoporphyria (EPP)
MeSH Terms: conditions — Protoporphyria, Erythropoietic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MT-7117 low dose (Experimental)
  Interventions: Drug: MT-7117 low dose
- MT-7117 high dose (Experimental)
  Interventions: Drug: MT-7117 high dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-7117 low dose — MT-7117 low dose QD, oral, 16 weeks
  Arms: MT-7117 low dose
Drug: MT-7117 high dose — MT-7117 high dose QD, oral, 16 weeks
  Arms: MT-7117 high dose
Drug: Placebo — Placebo QD, oral, 16 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of MT-7117 on sunlight exposure duration without symptoms and tolerance in subjects with EPP.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo controlled study to assess the efficacy, tolerability, and safety of MT-7117 in subjects with EPP. The study consists of a 2 week screening period, a 16 week double-blind treatment period, and a 6 week follow-up period at Week 22. The total participation period is approximately 24 weeks.

ELIGIBILITY:
Additional screening criteria check may apply for qualification.

Inclusion Criteria:

* 1. Subjects provided written informed consent to participate.
* 2. Male and female subjects with a confirmed diagnosis of EPP based on medical history, aged 18 years to 75 years, inclusive, at Screening.
* 3. Subjects are willing and able to travel to the study sites for all scheduled visits.
* 4. In the Investigator's opinion, subject is able to understand the nature of the study and any risks involved in participation, and willing to cooperate and comply with the protocol restrictions and requirements (including travel).

Exclusion Criteria:

* 1. History or presence of photodermatoses other than EPP.
* 2. Subjects who are unwilling or unable to go outside during daylight hours (e.g., between 1 hour post sunrise and 1 hour pre-sunset) during the study.
* 3. Presence of clinically significant hepatobiliary disease based on LFT values at Screening.
* 4. Subjects with AST, ALT, ALP ≥3.0 × upper limit of normal (ULN) or total bilirubin >1.5 × ULN at Screening.
* 5. Subjects with or having a history (in the last 2 years) of excessive alcohol intake in the opinion of the Investigator.
* 6. History or presence of melanoma and/or atypical nevus at Screening.
* 7. History of familial melanoma (defined as having 2 or more first-degree relatives, such as parents, sibling and/or child).
* 8. History or presence of pre-malignant skin lesion squamous cell carcinoma, basal cell carcinoma, or other malignant skin lesions.
* 9. History or presence of psychiatric disease judged to be clinically significant by the Investigator and which may interfere with the study evaluation and/or safety of the subjects.
* 10. Presence of clinically significant acute or chronic renal disease based upon the subject's medical records including hemodialysis; and a serum creatinine level of greater than 1.2 mg/dL or a glomerular filtration rate (GFR) <60 ml/min.
* 11. Presence of any clinically significant disease or laboratory abnormality which, in the opinion of the Investigator, can interfere with the study objectives and/or safety of the subjects.
* 12. Pregnancy or lactation.
* 13. Females of child bearing potential and male subjects with partners of child-bearing potential unwilling to use adequate contraception measures as described in the protocol.
* 14. Treatment with phototherapy within 3 months before Randomization (Visit 2).
* 15. Treatment with afamelanotide within 3 months before Randomization (Visit 2).
* 16. Treatment with cimetidine within 4 weeks before Randomization (Visit 2).
* 17. Treatment with antioxidant agents at doses which, in the opinion of the Investigator, may affect study endpoints (including but not limited to beta-carotene, cysteine, pyridoxine) within 4 weeks before Randomization (Visit 2).
* 18. Chronic treatment with prescription-based analgesic agents including but not limited to opioids and opioid derivatives such as morphine, hydrocodone, oxycodone or their combination with other analgesics or non-steroidal anti-inflammatory drug (NSAID, as Percocet and Vicodin-like prescription drugs) within 4 weeks before Randomization (Visit 2).
* 19. Treatment with any drugs or supplements which, in the opinion of the Investigator, can interfere with the objectives of the study or safety of the subjects.
* 20. Previous exposure to MT 7117.
* 21. Previous treatment with any investigational agent within 12 weeks before Screening OR 5 half-lives of the investigational product (whichever is longer).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-09-28 (Actual); Study Completion 2019-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (9):
- United States (9):
  - ACTCA, A Member of the Alliance, Inc., Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Metro Boston Clinical Partners, LLC, Brighton, Massachusetts
  - Ichan School of Medicine at Mount Sinai, New York, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Remington-Davis, Inc, Columbus, Ohio
  - University of Texas Medical Branch Porphyria Center, Galveston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Result] Balwani M, Bonkovsky HL, Levy C, Anderson KE, Bissell DM, Parker C, Takahashi F, Desnick RJ, Belongie K; Endeavor Investigators. Dersimelagon in Erythropoietic Protoporphyrias. N Engl J Med. 2023 Apr 13;388(15):1376-1385. doi: 10.1056/NEJMoa2208754. PMID 37043653
- [Derived] Ogasawara A, Ide R, Inoue S, Tsuda M, Teng R. Assessment of Potential Drug-Drug Interactions for Novel Oral Melanocortin-1 Receptor Agonist Dersimelagon. Pharmacol Res Perspect. 2025 Feb;13(1):e70069. doi: 10.1002/prp2.70069. PMID 39887900

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MT-7117 Low Dose | MT-7117 High Dose | Placebo
Started | 33 | 34 | 35
Completed | 31 | 30 | 31
Not Completed | 2 | 4 | 4
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 4
Not completed — CS Adverse Findings from Post- Baseline Nevi Evaluation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MT-7117 Low Dose | MT-7117 High Dose | Placebo | Total
Number analyzed (Participants) | 33 | 34 | 35 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (12.8) | 41.9 (14) | 38.1 (12.6) | 40.6 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 25 | 13 | 53
  Male | 18 | 9 | 22 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 32 | 32 | 34 | 98
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 33 | 33 | 32 | 98
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily Time (Minutes) to First Prodromal Symptom Associated With Sunlight Exposure Between Hour Post Sunrise and 1 Hour Pre-Sunset at Week 16.
Description: Duration in minutes, of sunlight exposure between 1 hour post sunrise and 1 hour pre-sunset. The average Duration in minutes, of sunlight exposure before the first prodromal symptom between 1 hour post sunrise and 1 hour pre-sunset. The average duration means that average of daily durations in 14-day windows before Day 1 (or week 16 Day) applied.
Time Frame: Baseline (Week 0) and Week 16
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | MT-7117 Low Dose | MT-7117 High Dose | Placebo
Number analyzed (Participants) | 33 | 34 | 35
Minutes | 74.7 (76.8) | 92.4 (100) | 21.0 (63.4)

2. Primary Outcome: Change From Baseline in Average Daily Duration (Minutes) of Sunlight Exposure Between 1 Hour Post Sunrise and 1 Hour Pre-Sunset Without Prodromal Symptoms at Week 16
Description: Change from baseline to week 16 in Average Daily Duration (Minutes) of Sunlight Exposure sums any sunlight exposure time excluding any overlapped time with prodromal symptoms, including if the patients go out multiple times on the same day after the prodromal symptom had previously ended.
Time Frame: Baseline (Week 0), and Week 16
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | MT-7117 Low Dose | MT-7117 High Dose | Placebo
Number analyzed (Participants) | 33 | 34 | 35
Minutes | 72.6 (76.2) | 86.1 (83.9) | 19.9 (63.2)

3. Primary Outcome: Change From Baseline in Average Daily Mean Duration (Minutes) of Sunlight Exposure Between 1 Hour Post Sunrise and 1 Hour Pre-Sunset Without Prodromal Symptoms at Week 16
Description: Change from baseline to week 16 in Average Daily Mean Duration (Minutes) of Sunlight Exposure without prodromal symptoms divided by the number of sunlight exposures periods applicable that day.
Time Frame: Baseline (Week 0), and Week 16
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | MT-7117 Low Dose | MT-7117 High Dose | Placebo
Number analyzed (Participants) | 33 | 34 | 35
Minutes | 70.2 (73.4) | 59.3 (85.2) | 12.8 (46.9)

4. Secondary Outcome: Total Number of Sunlight Exposure Episodes With Prodromal Symptoms During 16-Week Double-Blind Treatment Period
Time Frame: Week 16
Population: ITT Population
Measure: Mean (Standard Deviation); unit: sunlight exposure episodes
Arm/Group | MT-7117 Low Dose | MT-7117 High Dose | Placebo
Number analyzed (Participants) | 33 | 34 | 35
sunlight exposure episodes | 8.6 (9.3) | 7.7 (6.6) | 11.1 (13.3)

5. Secondary Outcome: Change From Baseline in Average Daily Mean Intensity of Prodromal Symptoms During 16-week Double-blind Treatment Period in 11-point Likert Scale
Description: The Intensity of Prodromal Symptoms is measured by 11-point Likert scale ranges from 0 (no symptom) to 10 (greatest severity of symptom).
Time Frame: Baseline (Week 0), and Week 16
Population: ITT Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MT-7117 Low Dose | MT-7117 High Dose | Placebo
Number analyzed (Participants) | 33 | 34 | 35
score on a scale
  Baseline: number analyzed (Participants) | 29 | 31 | 29
  Baseline | 2.0 (1.1) | 2.1 (0.9) | 2.0 (1.1)
  Week 16: number analyzed (Participants) | 8 | 7 | 12
  Week 16 | 1.7 (1.1) | 2.4 (1.7) | 2.4 (1.4)

6. Secondary Outcome: Change From Baseline in Average Daily Duration (Minutes) of Prodromal Symptoms at 16-Week Double-Blind Treatment Period
Time Frame: Baseline (Week 0), and Week 16
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | MT-7117 Low Dose | MT-7117 High Dose | Placebo
Number analyzed (Participants) | 33 | 34 | 35
Minutes | 55.3 (321.0) | 111.0 (466.1) | 83.3 (267.2)

7. Secondary Outcome: Change From Baseline in Pigmentation as Measured by Melanin Density for Average of 6 Skin Segments at Week 8 and Week 16.
Description: Pigmentation will be assessed in melanin density which are numeric scores measured by spectrophotometer on 6 skin segments (forehead, left cheek, right inside upper arm, left medial forearm, right-hand side of abdomen, and left-hand side of buttock).
Time Frame: Baseline (Week 0), Week 8, and Week 16
Population: ITT Population
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | MT-7117 Low Dose | MT-7117 High Dose | Placebo
Number analyzed (Participants) | 33 | 34 | 35
unitless
  Change from Baseline at Week 8: number analyzed (Participants) | 32 | 29 | 32
  Change from Baseline at Week 8 | 1.4635 (3.1644) | 1.6557 (2.2099) | 0.1390 (0.3376)
  Change from Baseline at Week 16: number analyzed (Participants) | 23 | 24 | 29
  Change from Baseline at Week 16 | 1.1413 (0.7285) | 1.5307 (0.6881) | 0.1639 (0.3939)

8. Secondary Outcome: Percent Change From Baseline in Pigmentation as Measured by Melanin Density for Average of 6 Skin Segments at Week 8 and Week 16.
Time Frame: Baseline (Week 0), Week 8, and Week 16
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | MT-7117 Low Dose | MT-7117 High Dose | Placebo
Number analyzed (Participants) | 33 | 34 | 35
percent change
  % Change from Baseline at Week 8: number analyzed (Participants) | 32 | 29 | 32
  % Change from Baseline at Week 8 | 30.4135 (32.8302) | 42.5543 (38.8390) | 4.2394 (11.9435)
  % Change from Baseline at Week 16: number analyzed (Participants) | 23 | 24 | 29
  % Change from Baseline at Week 16 | 44.0135 (43.7325) | 56.2871 (41.0660) | 7.4214 (16.7074)

9. Secondary Outcome: Total Number of Pain Events During 16-Week Double-Blind Treatment Period
Time Frame: Week 16
Population: ITT Population
Measure: Mean (Standard Deviation); unit: pain events
Arm/Group | MT-7117 Low Dose | MT-7117 High Dose | Placebo
Number analyzed (Participants) | 33 | 34 | 35
pain events | 4.0 (6.4) | 3.3 (2.8) | 5.4 (4.9)

10. Other Pre Specified Outcome: Total Number of Sunlight Exposure Episodes
Time Frame: Baseline (Week 0) and Week 16
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Pigmentation as Measured by Melanin Density
Time Frame: Baseline (Week 0) and Week 16
Reporting Status: Not Posted

12. Other Pre Specified Outcome: The Quality of Life as Measured by the Patient Reported Outcomes Measurement Information System (PROMIS) 57
Time Frame: Baseline (Week 0) and Week 16
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All AEs and SAEs that occurred from the time written informed consent was obtained until the end of the follow-up period (6 weeks after the last treatment visit, for safety monitoring)
Description: One subject who was randomized to Placebo received MT-7117 high Dose instead of placebo. Therefore, the subject was counted as MT-7117 high Dose Group in the Safety Population.
Arm/Group | MT-7117 Low Dose | MT-7117 High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 1/33 | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 31/33 | 34/35 | 31/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MT-7117 Low Dose (N=33) | MT-7117 High Dose (N=35) | Placebo (N=34)
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MT-7117 Low Dose (N=33) | MT-7117 High Dose (N=35) | Placebo (N=34)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Congenital naevus (Congenital, familial and genetic disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 5
Chapped lips (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 8 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 3
Nausea (Gastrointestinal disorders) | 5 | 16 | 4
Oral discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0
Pigmentation lip (Gastrointestinal disorders) | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3 | 1
Chest discomfort (General disorders) | 1 | 0 | 0
Chills (General disorders) | 1 | 2 | 0
Fatigue (General disorders) | 1 | 6 | 1
Pain (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 2 | 1
Ear infection (Infections and infestations) | 0 | 2 | 0
Folliculitis (Infections and infestations) | 1 | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0
Gastric infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 10 | 4 | 7
Sinusitis (Infections and infestations) | 0 | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 2 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chemical burn of skin (Injury, poisoning and procedural complications) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 2 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 3 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 7 | 3
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 3 | 0
Head discomfort (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 6 | 10 | 6
Paraesthesia (Nervous system disorders) | 1 | 2 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Actinic prurigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ephelides (Skin and subcutaneous tissue disorders) | 5 | 11 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Milia (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 5 | 5 | 3
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 3 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Sebaceous hyperplasia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 | 11 | 0
Solar dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Solar lentigo (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Yellow skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT03520036/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/36/NCT03520036/SAP_001.pdf